CLINICAL TRIAL: NCT04913116
Title: Agreement of Antigen Tests on Oral Pharyngeal Swabs or Less Invasive Testing With PCR, for Detecting SARS-CoV-2 in Adults: A Prospective Nationwide Observational Study
Brief Title: Generic Testing of Antigen Tests for COVID-19 in Denmark
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Herlev and Gentofte Hospital (Other); Odense University Hospital (Other); Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other); Slagelse Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Sygehus Lillebaelt (Other); Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Uffe Schneider, Principal Investigator., Hvidovre University Hospital
Other Study IDs: Nat COVID Ag Project
Record Dates: First submitted 2021-05-12; First posted 2021-06-04 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV2 Infection; COVID-19 Testing
Keywords: antigen test; RT-PCR; Prospective samples; Retrospective samples
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — SARS-CoV-2 samples are collected from SARS-CoV-2 positive and negative individuals, analyzed and discharged
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-Cov-2 positives: 200 individuals will be tested by each antigen test. Testing is done with up to three swabs at a time from each anatomical test location
  Interventions: Diagnostic Test: Comparison of antigen tests with RT-PCR as reference method
- SARS-CoV-2 negatives: 200 individuals will be tested by each antigen test. Testing is done with up to three swabs at a time from each anatomical test location
  Interventions: Diagnostic Test: Comparison of antigen tests with RT-PCR as reference method

INTERVENTIONS:
Diagnostic Test: Comparison of antigen tests with RT-PCR as reference method — Antigen tests are performed locally including sampling from multiple anatomical testing sites. A reference oropharyngeal swab is always send for RT-PCR for SARS-CoV-2 at DTU to verify the status of the patient. RT-PCR samples from other anatomical test locations may be included.

SUMMARY:
To evaluate the analytical and clinical sensitivity and specificity of antigen tests performed as oropharyngeal swabs, outer nasal swabs, saliva swabs or breath tests including self-tests for SARS-CoV-2 towards standard RT-PCR testing.

For each test 200 SARS-CoV-2 positive and 200 SARS-CoV-2 negative individuals previously defined by RT-PCR are tested. When tested an additional RT-PCR test is performed to verify status.

Analytical sensitivity and specificity is determined on 210 SARS-CoV-2 positive samples with known Cq and 100 SARS-CoV-2 negative samples.

30 companies with a total of 55 tests participate in this nationwide study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over,
* Capacity to give informed, written consent
* Be able to cooperate to the additional testing.

Exclusion Criteria:

* Individuals not fulfilling the inclusion criteria
* Declining additional oropharyngeal, nasal or saliva swabs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: approximately 4400 adult out-patients tested for SARS-CoV-2 by RT-PCR within 24 hours prior to inclusion.
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Clinical sensitivity and specificity of each antigen test compared to RT-PCR test result. | Up to 3 days after first initial positive COVI-19 RT-PCR test
  Performance is compared for each antigen test in relation to oropharyngeal RT-PCR samples collected simultaneously
Analytical sensitivity and specificity of each antigen test on retrospectively collected SARS-CoV-2 positive and negative samples. | 2 months
  SARS-CoV-2 positive samples are stratified into subgroups according to Cq by RT-PCR and frozen samples in universal transport medium is tested on each antigen test.

SECONDARY OUTCOMES:
Clinical sensitivity compared to RT-PCR result with the later stratified into low, intermediate and high Cq | Up to 3 days after first initial positive COVI-19 RT-PCR test
  Performance of each antigen test in relation to the cycle of quantification Cq by RT-PCR stratified into low (Cq <25), intermediate (Cq 25-35) and High (Cq >35).
Agreement between oropharyngeal swabs and tests from other anatomical test locations by RT-PCR. | Up to 3 days after first initial positive COVI-19 RT-PCR test.
  Antigen an RT-PCR tests are performed from multiple anatomical sampling sites on each teste individual.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Hvidovre University Hospital, Hvidovre
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Schneider UV, Knudsen JD, Koch A, Kirkby NS, Lisby JG. An Agreement of Antigen Tests on Oral Pharyngeal Swabs or Less Invasive Testing With Reverse Transcription Polymerase Chain Reaction for Detecting SARS-CoV-2 in Adults: Protocol for a Prospective Nationwide Observational Study. JMIR Res Protoc. 2022 May 4;11(5):e35706. doi: 10.2196/35706. PMID 35394449

DOCUMENTS (1):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT04913116/Prot_000.pdf